CLINICAL TRIAL: NCT05895409
Title: A Multicenter Prospective Study of Risk Factors in Progressive Pulmonary Fibrosis
Status: Recruiting | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Zhi Guo, Principal Investigator, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2023(029)
Record Dates: First submitted 2023-05-09; First posted 2023-06-08 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Interstitial Lung Disease
Keywords: progressive pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PF: Patients with interstitial lung disease (ILD) of known or unknown etiology other than IPF who has radiological evidence of pulmonary fibrosis(PF).

SUMMARY:
The goal of this observational study is to learn about risk of progressive pulmonary fibrosis (PPF). The main questions it aims to answer are:

* Risk factors of PPF
* Prevalence of PPF
* Mortality of PPF

Patients with interstitial lung disease (ILD) of known or unknown etiology other than IPF who has radiological evidence of pulmonary fibrosis will enroll in this study.

* All participants will have baseline investigations at the first visit having provided informed consent.
* At the first visit, baseline characteristics will be collected including demographics, medical history, smoking history, complications and medication use. 50 mL of blood will be obtained. High resolution computed tomography (HRCT), full lung function tests and a 6 min walk test will be performed.
* Further visits at 6 months and 12 months will include further 50 mL blood sampling. HRCT, full lung function tests and a 6 min walk test will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Agree and sign the informed consent form
* Interstitial lung disease patients with imaging features of pulmonary fibrosis

Exclusion Criteria:

* Patients with idiopathic pulmonary fibrosis (IPF)
* Pregnant or lactating women
* mental illness or cognitive impairment
* participating in other clinical studies
* Unable to sign informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the first affiliated Hospital of Shandong first Medical University,Jinan Central Hospital,Jinan people's Hospital,The fourth people's Hospital of Jinan and PLA 960 Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Establish the correlation between Age (years) and progression to PPF | Up to 12 months
Establish the correlation between Gender (the proportion of female and the proportion of male) and progression to PPF | Up to 12 months
Establish the correlation between Body mass index (BMI, kg/m2) and progression to PPF | Up to 12 months
Establish the correlation between ILD-Gender-Age-Physiology score (0-3,4-5 and 6-8) and progression to PPF | Up to 12 months
Establish the correlation between Artery blood gas and progression to PPF | Up to 12 months
  Artery blood gas: PaCO2 (mmHg) and PaO2 (mmHg)
Establish the correlation between Pulmonary function and progression to PPF | Up to 12 months
  Pulmonary function: forced vital capacity (FVC, L) and diffusion capacity for carbon monoxide of the lung (DLCO, mmol/min/kPa)
Establish the correlation between 6 min walk test distance (meters) and progression to PPF | Up to 12 months
Establish the correlation between Biomarkers and progression to PPF | Up to 12 months
  Biomarkers:CCL18(pg/mL),KL-6(pg/mL),CA125(pg/mL),MMP-7(pg/mL),SP-D(pg/mL) and IL-6(pg/mL)

SECONDARY OUTCOMES:
Prevalence of PPF | Up to 36 months
  Prevalence of PPF in patients with fibrosing ILD.

OTHER OUTCOMES:
Establish the correlation between Age (years) and mortality of PPF | Up to 36 months
Establish the correlation between Gender (the proportion of female and the proportion of male) and mortality of PPF | Up to 36 months
Establish the correlation between Body mass index (BMI, kg/m2) and mortality of PPF | Up to 36 months
Establish the correlation between ILD-Gender-Age-Physiology score (0-3,4-5 and 6-8) and mortality of PPF | Up to 36 months
Establish the correlation between Artery blood gas and mortality of PPF | Up to 36 months
  Artery blood gas: PaCO2 (mmHg) and PaO2 (mmHg)
Establish the correlation between Pulmonary function and mortality of PPF | Up to 36 months
  Pulmonary function: forced vital capacity (FVC, L) and diffusion capacity for carbon monoxide of the lung (DLCO, mmol/min/kPa)
Establish the correlation between 6 min walk test distance (meters) and mortality of PPF | Up to 36 months
Establish the correlation between Biomarkers and mortality of PPF | Up to 36 months
  Biomarkers:CCL18(pg/mL),KL-6(pg/mL),CA125(pg/mL),MMP-7(pg/mL),SP-D(pg/mL) and IL-6(pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China